CLINICAL TRIAL: NCT05648929
Title: Immunological Analysis of Capsular Tissue Formed Around Expanders With Varying Surface Topography in Women Undergoing Bilateral Nipple or Skin Sparing Mastectomy
Brief Title: Experimental and Clinical Investigation of the Implant Surface Roughness Reduction Effect on Early-stage Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EIT2020
Record Dates: First submitted 2022-11-10; First posted 2022-12-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-01

CONDITIONS: Capsular Contracture Associated With Implant; Foreign-Body Reaction; Wounds and Injuries; Tissue Expander Disorder
Keywords: prophylactic NSME (nipple sparing mastectomy); implant-based breast reconstruction; medical grade silicone; SMI (silicone mammary implants); Foreign body response to SMI; SMI encapsulation; immunoreactivity of SMI surface topography; capsular fibrosis; immunomodulation by SMI-surface roughness
MeSH Terms: conditions — Foreign-Body Reaction; Wounds and Injuries | interventions — Pregnancy Tests; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: intraindividual comparative analysis of two different devices implanted within one individual patient.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: randomised double-blinded trial: A total of 14 patients will receive either Motiva SmoothSilk® or other routinely used expander (Mentor CPX™4) randomized to left or right breast after mastectomy. Patient and laboratory expert will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the conventional expander Mentor CPX4 (MENTOR) (Active Comparator): intraindividual comparison of two differentially rough tissue expanders
  Arm description: women undergoing prophylactic bilateral NSME and simultaneous tissue-expander based reconstruction with conventionally textured expander with surface roughness 60µM Ra
  Interventions: Other: Patient Satisfaction Questionnaire; Diagnostic Test: Pregnancy test; Procedure: Blood draw; Procedure: Expander based breast reconstruction; Procedure: Ultrasound of breast; Other: S(AE )monitoring
- the expander SmoothSilk(Motiva) with reduced surface roughness (Active Comparator): intraindividual comparison of two differentially rough tissue expanders
  Arm description: women undergoing prophylactic bilateral NSME and simultaneous tissue-expander based reconstruction with reduced textured expander with surface roughness 4µM Ra
  Interventions: Other: Patient Satisfaction Questionnaire; Diagnostic Test: Pregnancy test; Procedure: Blood draw; Procedure: Expander based breast reconstruction; Procedure: Ultrasound of breast; Other: S(AE )monitoring

INTERVENTIONS:
Other: Patient Satisfaction Questionnaire — During regular clinical examinations patient will go through a short questionnaire at week 4, 16 and 24 to check patient satisfaction with expanders
Diagnostic Test: Pregnancy test — Pre-op; to sufficiently check pregnancy as exclusion criteria
Procedure: Blood draw — pre- expander implantation, alongside anaesthesia pre- expander explantation and exchange with definite implant alongside anaesthesia - no additional vein irritation needed
Procedure: Expander based breast reconstruction — implantation of 2 different expanders intraindividually
Procedure: Ultrasound of breast — Measurement of capsular thickness pre- expander removal
Other: S(AE )monitoring — (S)AE evaluation will be performed from Visit 1 (Day 0 = Expander implantation) to Visit 15 (Day 168-196 = Reoperation) according to visit plan.

SUMMARY:
The goal of this single-center, randomised double-blinded trial is to compare the early stage fibrosis progression around conventional textured expander and the SmoothSilk® expander with reduced surface roughness in women undergoing bilateral nipple or skin sparing mastectomy in a prophylactic setting followed by tissue-expander based breast reconstruction. Researchers will compare intra-individually, the conventional textured expander CPX®(Mentor) and the SmoothSilk® (Motiva) expander (i) to gain a comprehensive insight into immunological mechanisms occurring at the timepoint of expander insertion (within the first days after implantation) based on WBF analysis in vitro, (ii)to determine the role and function of immune cells in a rather early stage of capsule formation (6-8 months after implantation) and under well-defined conditions in humans as well as (iii)to analyze the aesthetic outcome and clinical parameters after bilateral implant-based reconstruction using two expanders with varying surface topography within the individual patient (intra-individually).

DETAILED DESCRIPTION:
Expander Immunology trial is a single-center, randomized double-blinded trial. A total of 14 patients, undergoing prophylactic bilateral simultaneous NSME (nipple sparing mastectomy) and implant based breast reconstruction, will receive either SmoothSilk® (Motiva Flora) or other routinely used expander (Mentor CPX™4), randomised to left or right breast after mastectomy. Patient and laboratory expert will be double-blinded. Clinical follow-up visits will be scheduled at 2, 4, 5, 6, 7, 8 and 16 weeks post procedure. Biological sample collection of wound bed fluid will take place daily from day 1 to 5 after expander implantation. Ultrasound will be performed -28 to-1 day before re-operation. Capsule tissue will be harvested and blood draw will be performed during re-operation between 24 to 28 weeks after initial expander implantation.

Directly postoperatively at day 1-5 after expander implantation, wound bed fluid will be collected and proteinaceous and cellular components will be analyzed via FACS (flow cytometry), molecular (RNA, protein) assays and microbiome testing platform.

Phenotypical and functional analyses will be performed for capsular tissue and blood as well as PCR (polymerase chain reaction) assays for bacterial antigens when expanders are changed to definite implants. Expanders will also undergo sonication to check for bacterial contamination. Peri-capsular tissue samples will be evaluated using scanning electron microscopy-energy dispersive x-ray spectroscopy (SEM-EDS) to identify sites with/without titanium particles (Titan-Bra debris). And breast ultrasound will be performed to detect capsular thickness before the reoperation.

During regular clinical examinations patients will go through a short questionnaire at week 4 and 16 to check patient satisfaction with expanders and adverse events will be monitored. (S)AE evaluation will be performed from Visit 1 (Day 0 = Expander implantation) to Visit 15 (Day 168-196 = Reoperation) according to visit plan.

The main question[s] it aims to answer are:

1. Does the immune cell profile differ within the wound-bed fluid (WBF) directly after implantation? Do the investigators see different activation patterns or distribution patterns of immune cells within the WBF on the conventional expander reconstructed side versus the SmoothSilk® (Motiva) reconstructed side?
2. Does the immune cell profile differ within the capsular tissue formed around conventional expanders versus SmoothSilk® (Motiva) expanders?
3. Which cytokines are mainly expressed in the early capsular tissue (conventional expander versus SmoothSilk® (Motiva) and do the investigators see differences in comparison with those of peripheral blood?
4. Does the cellular composition (histology) show different distribution patterns of immune cells and ECM proteins in these capsules?
5. Do the investigators see differences concerning bacterial & fungi contamination in WBF and on expander shells at the time point of explantation (sonication and PCR as well as next-generation DNA sequencing for bacteria and fungi)
6. Do the investigators see titanium wear particle incorporation into peri-capsular tissue? Is there a difference between the conventional expanders versus SmoothSilk® (Motiva) expanders after 6-8 months?
7. Do the investigators see any differences in outcome analysis between the conventional expanders versus Motiva nano-textured expanders after 6-8 months (Seroma formation, Implant dislocation, thickness of capsule)?

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Female sex
* High risk family history for mammary and/or ovarian cancer
* Planned prophylactic mastectomy with simultaneous breast reconstruction
* Signed informed consent form

Exclusion Criteria:

* Confirmed sever Coagulation disorder, representing a potential contraindication for the elective surgery
* Confirmed Rheumatic disease accompanied by obligatory intake of immunomodulating therapeutic agents
* Confirmed severe renal functional disorder: Renal insufficiency status IV or V
* Active hematological or oncological disease
* HIV-Infection
* Hepatitis-Infection
* Pregnancy or breast feeding
* Intake of anti-inflammatory drugs
* Carrier of silicone implants (e.g. gastric banding, mammary implants)
* Subject is currently participating or intends to participate in another clinical trial that may interfere with the protocol of this study
* Patients who have implanted devices that could be affected by a magnetic field (e.g., pacemakers, drug infusion devices, artificial sensing devices) * patients with removable devices such as removable diabetes pumps, sensors and transmitter might still part take,
* Patients with alteration in hematologic and serum protein reference values post-chemotherapy.
* When there is a residual malignancy in the intended expansion site.
* Existing tissue at the intended expansion site is not adequate according to the surgeon's criteria, because of previous radiation therapy, ulcerations, vascular compromise, history of compromised wound healing, or scar deformity.
* Radiation therapy before or after the expander placement can be associated with a higher rate of complications during the expansion and final implantation phases of the reconstructive process.
* Abscess or infection in the body in general.
* Participants with autoimmune diseases (e.g., lupus, scleroderma) or whose immune system is compromised (e.g., currently receiving immunosuppressive therapy such as steroids).
* Unsuitable tissue due to radiation damage on the chest wall, tight thoracic skin grafts or radical resection of the pectoralis major muscle.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
wound bed fluid Immune cell profile (composition) | 1 to 5 days post expander implantation
  immediately after implantation wound drain fluid will be immune profiled for cell populations by flow cytometry to gain a comprehensive insight into immunological mechanisms occurring at the time-point of expander insertion (within the first days after implantation) and evaluate potential effects of expander surface roughness
wound bed fluid wound proteome composition | 1 to 5 days post expander implantation
  immediately after implantation wound drain fluid will be proteomically profiled by Mass Spectrometry for tissue repair and foreign body response to gain a comprehensive insight into immunological triggers and mechanisms occurring at the time-point of expander insertion (within the first days after implantation) and evaluate potential effects of expander surface roughness
wound bed fluid Immune cell activity | 1 to 5 days post expander implantation
  immediately after implantation wound drain fluid will be immune profiled for cell activity by qPCR analysis of cytokine expression to gain a comprehensive insight into immunological mechanisms occurring at the time-point of expander insertion (within the first days after implantation) and evaluate potential effects of expander surface roughness
wound bed fluid wound microbiome composition | 1 to 5 days post expander implantation
  will be NextGen sequenced for microbiome colonisation, population, and biofilm formation to gain a comprehensive insight into immunological triggers and mechanisms occurring at the time-point of expander insertion (within the first days after implantation) and evaluate potential effects of expander surface roughness

SECONDARY OUTCOMES:
Intracapsular immune cell composition | At reoperation; 6-8 months post expander implantation
  After 6-8 months, collected capsular tissue formed around both expanders will be analyzed for immune cell profile and composition by flow cytometry
Clinical evaluation of aesthetic outcome and postoperative complications | 2, 4 and 16 weeks and at reoperation; 6-8 months post expander implantation
  In follow-up visits 2, 4, and 16 W post-expander implantation; Breast will be clinically evaluated for symmetry and complications through clinical evaluation by the senior surgeon.
Intracapsular immune cell activity | At reoperation; 6-8 months post expander implantation
  After 6-8 months, collected capsular tissue formed around both expanders will be analyzed for immune cell activity and cytokine secretion and expression by qPCR
Ultrasound evaluation of capsular thickness and postoperative complications | At reoperation; 6-8 months post expander implantation
  Directly before the expanders are exchanged (6-8 months post implantation), an experienced radiologist will perform non-invasive ultrasound evaluation of capsular thickness and seroma formation.At last cosmetic outcome will be evaluated (breast symmetry, nipple areola complex).
Expander Satisfaction and comfortability evaluation by Questionnaire | At reoperation; 6-8 months post expander implantation
  Directly before the expanders are exchanged (6-8 months post implantation),, and expander comfortability as well as practicability during filling and expansion will be evaluated by the patient and senior surgeon on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Wolfram-Raunicher, Dr., Principal Investigator — Medical University of Innsbruck, Department for Plastic Surgery
Locations (1):
- Medical University of Innsbruck, Department for Plastic, Aethetic and Reconstructive Surgery, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
The sponsor Medical University Innsbruck and Principal investigator Assoc. Prof. PD. Dr. Wolfram intent to publish the results of this clinical investigation. The ownership of the data shall at all times be held by Medical University Innsbruck and the PI, who will be the main author of all publications by this trial.
  For the avoidance of doubt, positive and negative results may be published.

REFERENCES:
- [Result] Schoberleitner I, Augustin A, Egle D, Brunner C, Amort B, Zelger B, Brunner A, Wolfram D. Is It All about Surface Topography? An Intra-Individual Clinical Outcome Analysis of Two Different Implant Surfaces in Breast Reconstruction. J Clin Med. 2023 Feb 7;12(4):1315. doi: 10.3390/jcm12041315. PMID 36835850
- [Result] Schoberleitner I, Faserl K, Sarg B, Egle D, Brunner C, Wolfram D. Quantitative Proteomic Characterization of Foreign Body Response towards Silicone Breast Implants Identifies Chronological Disease-Relevant Biomarker Dynamics. Biomolecules. 2023 Feb 6;13(2):305. doi: 10.3390/biom13020305. PMID 36830674
- See also: Results reference — https://www.frontiersin.org/journals/immunology/articles/10.3389/fimmu.2024.1342895/abstract